CLINICAL TRIAL: NCT06551337
Title: Prospective Clinical Study on Vitamin D Replacement in Bronchiectasis - A Pilot Study
Brief Title: Vitamin D Replacement in Bronchiectasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Wang Chun, Clinical Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 24-205
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: 104 subjects will be separated into two groups according to their Baseline blood 25-hydroxyvitamin-D level: vitamin D deficient (below 50 nmol/L) and vitamin D non-deficient (at or above 50 nmol/L). There were initially 42 and 62 patients in the vitamin D deficient and vitamin D non-deficient groups respectively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D replacement (Active Comparator): Those with vitamin D deficiency will be replaced with vitamin D3 at 1000 IU at the first visit. Vitamin D3 1000 IU is expected to increase blood 25-hydroxyvitamin-D level by 25 nmol/L. Blood 25-hydroxyvitamin-D level will be rechecked 3 months after replacement. If the blood 25-hydroxyvitamin-D level is still below 50 nmol/L, the vitamin D3 replacement dosage will be increased to 2000 IU.
  Interventions: Drug: Vitamin D3
- Vitamin D non-deficiency (No Intervention): No drug will be given to patients with Vitamin D non-deficiency.

INTERVENTIONS:
Drug: Vitamin D3 — The non-CF bronchiectasis subjects with Vitamin D deficiency would be given 1000 IU and 2000 IU.
  Arms: Vitamin D replacement

SUMMARY:
This study seeks to address the limitations in previous related studies on vitamin D replacement and bronchiectasis exacerbation occurrence through a self-controlled pilot study. The investigators aim to investigate whether vitamin D replacement in bronchiectasis patients with vitamin D deficiency can reduce hospitalized bronchiectasis exacerbation occurrence. Patients who participated in the prior study entitled "Prospective clinical study on serum 25-hydroxyvitamin D (25-OH D) level and risk of bronchiectasis exacerbation" (UW 22-317) will be invited for participation during regular clinic follow-up and management in Queen Mary Hospital. If participants are willing to join the further research, participants will be recruited in this self-controlled study. There are some differences from usual management to non-CF bronchiectasis subjects. The study subjects would be checked for their blood 25-hydroxyvitamin-D level during the study period. The non-CF bronchiectasis subjects with Vitamin D deficiency would be given 1000 IU and 2000 IU (if needed). The investigators aim to correct their Vitamin D deficiency completely, aiming at blood 25-hydroxyvitamin-D level >=50, i.e. treat to target. The dose depends on the level of Vitamin D after replacement. If blood 25-hydroxyvitamin-D level is 50 or above, then 1000 IU is suffice. If blood 25-hydroxyvitamin-D level is still below 50, the investigators will increase to 2000 IU.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18 years or above, male or female.
2. confirmed diagnosis of non-CF bronchiectasis based on high-resolution computed tomography (HRCT) scan.
3. participation in the prior study entitled "Prospective clinical study on serum 25-hydroxyvitamin D (25-OH D) level and risk of bronchiectasis exacerbation" (UW 22-317)

Exclusion Criteria:

1. underlying asthma, COPD and other co-existing respiratory diseases
2. underlying osteoporosis
3. supplementary Vitamin D in their regimen
4. advanced chronic kidney disease with estimated glomerular filtration rate (eGFR) < 30mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who develop hospitalized bronchiectasis exacerbation | From 1-year period before baseline to 12 months
  The proportion of patients who develop hospitalized bronchiectasis exacerbation during the follow-up period of 12 months, when compared with the 1-year period before.

SECONDARY OUTCOMES:
Change in St. George's Respiratory Questionnaire (SGRQ) score | From baseline to 6 and 12 months.
  Scores range from 0 to 100, with higher scores indicating more limitations.
Change in bronchiectasis impact measure (BIM) score | From baseline to 6 and 12 months.
  A score ranges from 0 to 10 for each of eight domains consists of cough, sputum, breathlessness, tiredness, activity, general health, control, and exacerbation, with 10 being most severe.
Change in Bronchiectasis Health Questionnaire (BHQ) score | From baseline to 6 and 12 months.
  The instrument comprises 10 questions, each scored on a 7-point scale, to assess quality of life related to bronchiectasis on individuals for a recall period of 2 weeks. The total score ranges from 10 to 70, with a lower score indicating a more negative impact on health-related quality of life (HRQOL).

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT06551337/Prot_000.pdf
  • Informed Consent Form (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT06551337/ICF_001.pdf